CLINICAL TRIAL: NCT06361680
Title: Efficacy of Coenzyme Q10 Supplementation on Metabolic Control in Children With Type 1 Diabetes Mellitus: a Randomized Clinical Trial
Brief Title: Effect of Coenzyme Q10 on Diabetic Children
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Christina Saad Abdel Malak Abdel Nour, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Coenzyme Q10 on diabetic child
Record Dates: First submitted 2024-03-15; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Will take Coenzyme Q10 soft gel capsules or tablets in a dose of 100-200mg of natural factors
  Interventions: Drug: Coenzyme Q10 Cap/Tab as natural factors capsules or kirkman tablets
- Group B (Experimental): Will not take Coenzyme Q10 soft gel capsules or tablets
  Interventions: Drug: Coenzyme Q10 Cap/Tab as natural factors capsules or kirkman tablets

INTERVENTIONS:
Drug: Coenzyme Q10 Cap/Tab as natural factors capsules or kirkman tablets — Group A will take Soft gel capsules or tablets of Coenzyme Q10 in a dose of 100-200mg of natural factors or kirkman but group B will not take Coenzyme Q10 just observe them
  Other Names: Natural factors capsules or Kirkman tablets

SUMMARY:
Determine the effect of Coenzyme Q10 on random blood sugar and glycosylated haemoglobin

DETAILED DESCRIPTION:
Type 1 diabetes mellitus is an autoimmune disease that leads to destruction of insulin producing pancreatic Beta cells.

Individuals with type 1 diabetes requires life long insulin replacement with multiple daily insulin injection. daily,insulin pump therapy or the use of an automated insulin delivery system.

without insulin ,diabetic ketoacidosis develops and is life threatening.

In addition to insulin Therapy ,glucose monitoring with a continuous glucose monitor and a blood glucose monitor if continuous glucose monitor is unavailable is recommended .

Coenzyme Q10 supplementation has beneficial effects on glycemic control especially in diabetes , and 100-200 mg per day of Co Q10 could achieve the greatest benefit which could provide a basis for the dietary guidelines of Co Q10 in patients with glycemic disorders .

Co Q10 with a known antiinflammatory and antioxidant has beneficial effects on endothelial function and therefore minimize the microvascular and macrovascular complication in patients with type 1 diabetes mellitus.

Administration of Co Q10 for 3 months in type 1 diabetes mellitus in pediatric patients was will tolerated but had no favorable effect on endothelial dysfunction or metabolic parameters .

Co Q10 in addition to improving the metabolic hyperglycemia , it improve Hb A1c and the lipid profile.

patients with type 1 diabetes , especially poorly controlled had elevation of plasma vitamin E and coenzyme Q10 levels and decreased platelet redox status of coenzyme Q10 which may be an indicator of increased oxidative stress ,so Co Q10 has an antioxidant effects.

Researches on this topic are limited on pediatrics and investigators search for it and will see the result.(clinical trial)

Co Q10 is present in the forms of soft gel capsules ,oral spray , hard gel capsules and tablets .

Co Q10 approved from age of 2 years old to 18 years old .

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed as type 1 diabetes mellitus from age of 2 years old to 18 years old with diabetes mellitus of duration at least 1 year.

Exclusion Criteria:

* - patients diagnosed as diabetes mellitus less than 2 years old .
* patients with diabetes mellitus of duration less than 1 year.
* patients diagnosed as type 1 diabetes mellitus with Thyroid or celiac diseases.
* other types of hyperglycemia rather than Type 1 diabetes mellitus.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Assess the effect of Coenzyme Q10 on glycated haemoglobin in type 1 diabetes mellitus | One year
  This prospective randomized clinical trial will be conducted on 100 participants . Half of them will not receive treatment but group A will receive 100-200mg of Coenzyme Q10 . the level of glycated hemoglobin, fasting blood glucose will be assessed for both groups at baseline and after 3 months of treatment for ongoing use in diabetic children

SECONDARY OUTCOMES:
Control of random blood sugar and glycated haemoglobin in children with type 1 diabetes mellitus . | One year
  By ensuring of regular intake of Coenzyme Q10 capsules or tablets then assessment of glycated hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Christina Saad Abdel Malak Abdel Nour, Principal Investigator — Study producer

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serag H, El Wakeel L, Adly A. Coenzyme Q10 administration has no effect on sICAM-1 and metabolic parameters of pediatrics with type 1 diabetes mellitus. Int J Vitam Nutr Res. 2021 Jun;91(3-4):315-324. doi: 10.1024/0300-9831/a000636. Epub 2020 Jan 16. PMID 31942840
- [Background] Sangouni AA, Taghdir M, Mirahmadi J, Sepandi M, Parastouei K. Effects of curcumin and/or coenzyme Q10 supplementation on metabolic control in subjects with metabolic syndrome: a randomized clinical trial. Nutr J. 2022 Oct 3;21(1):62. doi: 10.1186/s12937-022-00816-7. PMID 36192751
- [Background] Liang Y, Zhao D, Ji Q, Liu M, Dai S, Hou S, Liu Z, Mao Y, Tian Z, Yang Y. Effects of coenzyme Q10 supplementation on glycemic control: A GRADE-assessed systematic review and dose-response meta-analysis of randomized controlled trials. EClinicalMedicine. 2022 Aug 3;52:101602. doi: 10.1016/j.eclinm.2022.101602. eCollection 2022 Oct. PMID 35958521
- [Background] Stojanovic M, Radenkovic M. A meta-analysis of randomized and placebo-controlled clinical trials suggests that coenzyme Q10 at low dose improves glucose and HbA1c levels. Nutr Res. 2017 Feb;38:1-12. doi: 10.1016/j.nutres.2016.12.001. Epub 2016 Dec 8. PMID 28381349
- [Background] Salardi S, Zucchini S, Elleri D, Grossi G, Bargossi AM, Gualandi S, Santoni R, Cicognani A, Cacciari E. High glucose levels induce an increase in membrane antioxidants, in terms of vitamin E and coenzyme Q10, in children and adolescents with type 1 diabetes. Diabetes Care. 2004 Feb;27(2):630-1. doi: 10.2337/diacare.27.2.630. No abstract available. PMID 14747266